CLINICAL TRIAL: NCT01095822
Title: A Randomized Evaluation of the Effects of Valsartan and Aliskiren in Combination Versus Tekturna Alone on Hemostatic Biomarkers in Patients With Newly Diagnosed Mild to Moderate Hypertension and Type 2 Diabetes Mellitus
Brief Title: Effects of Valsartan and Aliskiren on Hemostatic Indices in Hypertensive Diabetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: HeartDrug Research LLC (Other)
Collaborators: Novartis (Industry)
Responsible Party: Victor Serebruany, HeartDrug Research LLC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DT-NOV-09-37918
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Last update posted 2010-03-30 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Hypertension; Platelets; Hemostasis; Aliskiren; Valsartan
MeSH Terms: conditions — Diabetes Mellitus; Hypertension | interventions — aliskiren; Valsartan

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aliskiren (Active Comparator): 25 patients with recently diagnosed hypertension and mild to moderate type 2 diabetes will constitute the proposed study population. The diagnosis of diabetes will be made based on the American Diabetes Association criteria, such as random plasma glucose >200 mg/dL with or without symptoms of hyperglycemia (polydipsia, polyuria, polyphagia) and weight loss, or fasting plasma glucose > 126 mg/dL, to be determined at least twice. Patients will qualify if they are insulin-free, treated with an oral antiglycemic agent,(metformin only) and/or managed on diet alone for no less than 30 days and have adequate glucose control at the time of their Screening Visit.
  Interventions: Drug: Aliskiren + Valsartan
- Aliskiren + Valsartan (Experimental): 25 patients with recently diagnosed hypertension, and mild to moderate type 2 diabetes will constitute the proposed study population. The diagnosis of diabetes will be made based on the American Diabetes Association criteria, such as random plasma glucose >200 mg/dL with or without symptoms of hyperglycemia (polydipsia, polyuria, polyphagia) and weight loss, or fasting plasma glucose > 126 mg/dL, to be determined at least twice. Patients will qualify if they are insulin-free, treated with an oral antiglycemic agent,(metformin only) and/or managed on diet alone for no less than 30 days and have adequate glucose control at the time of their Screening Visit.
  Interventions: Drug: Aliskiren + Valsartan

INTERVENTIONS:
Drug: Aliskiren + Valsartan — Comparison of combination (aliskiren + valsartan) therapy versus valsartan alone on hemostatic indices

SUMMARY:
People with both hypertension and diabetes have a higher chance of developing heart and arterial problems that could be reduced with anti-coagulant therapy. Valsartan (Diovan), an FDA approved angiotensin-II receptor antagonist (blocker) clinically indicated for the treatment of essential hypertension is known to inhibit platelet activity in both an in vitro and ex vivo setting. Aliskiren (Tekturna) is a recently FDA-approved potent direct renin inhibitor which is also an effective anti-hypertensive agent in patients with mild-to-moderate hypertension and which, in vitro, modulates antithrombin III in plasma. Therefore, in addition to being clinically approved anti-hypertensive medications, combining these two agents will potentially target both primary hemostasis (platelets) and anticoagulant (antithrombin-III is a cornerstone substrate for heparin) properties to exert their anti-thrombotic efficacy simultaneously. This combination strategy may not only improve hypertension management, but also improve vascular outcomes in high-risk diabetic population via favorable effects on anti-thrombotic activity. Importantly, there have been no significant additional safety concerns of using the combination of aliskiren and valsartan. The investigators hypothesis is that valsartan 160 mg/daily in combination with aliskiren 150-300 mg/daily for 4 weeks will favorably affect blood levels of platelet/coagulation/fibrinolytic biomarkers (ie, diminish platelet activity, and enhance antithrombin III potency) when compared with monotherapy with aliskiren 150mg/daily in hypertensive patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Objectives:

There are 2 objectives in the index study. • The primary objective is to determine how therapy with valsartan (160mg/daily) in combination with aliskiren (150-300mg/daily) over four weeks affects platelet/coagulation/fibrinolytic biomarkers in recently diagnosed hypertensive patients with type 2 diabetes mellitus. However, this is an exploratory study, our current knowledge is based on in vitro and ex vivo evidence for valsartan, but only on in vitro aliskiren data. There are no data on antithrombotic biomarkers currently available for the combination therapy.

The secondary objective is:

• To define whether combination therapy is superior over monotherapy with aliskiren with regard to the improvement of hemostatic biomarkers (platelet aggregation, expression of GP IIb/IIIa, and plasma levels of antithrombin-III).

Study Design:

This is a randomized 1:1, two arm, single-blind, single-site, parallel group, post-marketing comparison study of the effects on antithrombotic biomarkers of aliskiren 150-300mg/day alone vs combined treatment with aliskiren 150-300mg/day plus valsartan 160mg/day over a four week primary treatment period. An optional four week extension phase may be offered pending assessment of the antithrombotic biomarker assays at week four.

Population:

Two groups (25 patients each), for a total of 50, recently diagnosed hypertensive patients with previously diagnosed mild to moderate type 2 diabetes will constitute the proposed study population. The diagnosis of diabetes will be made based on the American Diabetes Association criteria, such as random plasma glucose >200 mg/dL with or without symptoms of hyperglycemia (polydipsia, polyuria, polyphagia) and weight loss, or fasting plasma glucose > 126 mg/dL, to be determined at least twice. Patients will qualify if they are insulin-free, treated with an oral antiglycemic agent,(metformin only) and/or managed on diet alone for no less than 30 days and have adequate glucose control at the time of their Screening Visit.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of Type 2 Diabetes Mellitus will have been determined by the following Criteria, as characterized by recurrent or persistent hyperglycemia, and diagnosed by demonstrating any one of the following.

   * Fasting plasma glucose level at or above 126 mg/dL but less than 250 mg/dL on more than one determination.
   * Plasma glucose at or above 200 mg/dL two hours after a 75 g oral glucose load as in a glucose tolerance test.
   * Symptoms of hyperglycemia and casual plasma glucose at or above 200 mg/dL.
   * Glycated hemoglobin (hemoglobin A1C) at or above 6.5 but below 8.5%. (This criterion was recommended by the American Diabetes Association in 2010).
2. Adults between 21 - 65 years old
3. Have been diagnosed with Type 2 DM according to the criteria listed above, and treated with metformin 1-2 g/daily as their only diabetic medication, and/or an approved ADA diet for no less than 30 days.
4. Documented evidence of Stage 1 or Stage 2 essential hypertension as noted below: However, the actual treatment threshold will be left to the discretion of the study investigators.

   Stage 1: systolic 140-159 mmHg and diastolic 90-99 mmHg Stage 2: systolic >160 mmHg and diastolic >100 mmHg However, there is accumulated evidence that patients with consistent blood pressures over 130/80 mmHg along with Type 1 or Type 2 diabetes, or kidney disease are at increased risk for progressive morbidity and mortality and require a lower threshold for further treatment.
5. Aspirin 81 mg/daily
6. Signed informed consent
7. Must maintain same diet/exercise regimen

Exclusion Criteria:

1. Thrombolytic therapy, GP IIb/IIIa inhibitor, thienopyridines, antifibrinolytics, COX- inhibitors, prostacyclin analogues, and vitamin K antagonists within 30 days of enrollment
2. Platelet count < 100,000/microL
3. History of bleeding disorder
4. Hct < 30%, serum creatinine ≥3 mg/dL, liver impairment defined as ALT/AST > 3 times upper limit of normal.
5. Glomerular filtration rate <60ml/min/1.73m2
6. Patients currently treated with any antiplatelet agent other than aspirin 81 mg/day
7. Admission for acute vascular syndrome (unstable angina, MI, stroke), revascularization procedure with stent placement, or other major coronary/cerebrovascular event within 30 days.
8. Active participation in other investigational drug or device trial within the last 30 days.
9. Allergy or intolerance to any of the study medications.
10. Congestive Heart Failure (NYHA I-IV)
11. Malignancies except treated non-melanoma superficial skin cancers
12. Acute infections
13. Type I diabetes, Cushings syndrome, or pancreatic deficiency due to malignancy or systemic disease
14. Insulin therapy, sulfonylureas, thiazolidinediones,meglitinides, D-phenylalanine derivatives, amylin synthetic derivatives, and incretin mimetics.
15. Pregnancy, confirmed by serum rosette inhibition assay for early pregnancy factor detectable. For women of child-bearing potential (WOCP), continuous abstinence, fertility awareness, hormonal contraceptives, and/or mechanical methods will apply to prevent pregnancy during the entire study duration. Should a subject become pregnant during the study, the anti-hypertensive treatment with either or both study medications will be discontinued immediately by the treating physician/investigator as per FDA warnings regarding potential fetal/neonatal morbidity and mortality.
16. Age over 65 years
17. History of cigarette smoking within past 10 years

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
How therapy with valsartan (160mg/daily) in combination with aliskiren (150-300mg/daily) affects platelet/coagulation/fibrinolytic biomarkers in recently diagnosed hypertensive patients with type 2 diabetes mellitus. | 4 weeks

SECONDARY OUTCOMES:
Whether combination therapy is superior over monotherapy with aliskiren with regard to the improvement of hemostatic biomarkers (platelet aggregation, expression of GP IIb/IIIa, and plasma levels of antithrombin-III). | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victor Serebruany, MD, PhD, Study Director — HeartDrug Research LLC
Locations (1):
- Dr. Pokov's Polyclinic. 6821 Reisterstown Road Suite 206, Baltimore, Maryland, United States

REFERENCES:
- See also: Core laboratory facility — http://www.heartdrug.com